CLINICAL TRIAL: NCT04992403
Title: Ocular Biometric Measurements in Cataract Surgery Candidates in The South of France : a Multicenter Cross Sectional Study
Brief Title: Ocular Biometrics in a French Population
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0458
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Cataract
Keywords: Biometry; Axial length; Cataract; Gender; High myopia
MeSH Terms: conditions — Cataract; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to study ocular biometrics parameters and their association with age, gender and the prevalence of high myopia in a population of cataract surgery candidates in the South of France. The investigators also aimed to define proportion of an "usual eye" and know the rate of inhomogeneous eyes in our population.

ELIGIBILITY:
Inclusion criteria:

* aged 40 years
* olderpatients who underwent ocular biometrics before cataract surgery

Exclusion criteria: incomplete examination

* previous cataract surgery
* age < 40 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent ocular biometrics before cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 11650 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
number of patients with Distribution of ocular biometrics | 1 day
  Distribution of ocular biometrics and their association with age and gender

SECONDARY OUTCOMES:
number of patients with Prevalence of high myopia | 1 day
  Prevalence of high myopia
rate of inhomogeneous eyes | 1 day
  rate of inhomogeneous eyes

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DAIEN, MD, PhD, HDR, Study Director — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC